CLINICAL TRIAL: NCT03106012
Title: The Value of Diagnostic Hysterolaparoscopy in Infertile Patients With Normal Hysterosalpingography
Brief Title: The Role of Hysterolaparoscopy in Infertile Patients With Normal Hysterosalpingography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 163
Record Dates: First submitted 2017-03-19; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Hysteroscopy; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hsyterolaparoscopy (Experimental): Subjected to bath diagnostic hystroscopy and laparoscopy
  Interventions: Procedure: Hysteroscopy; Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Hysteroscopy — rigid continuous flow diagnostic hysteroscopy (Tuttligen, Karl Storz, Germany). It has a 30o panoramic optic which is 4mm in diameter and the diagnostic continuous flow outer sheath is 6.5 mm in diameter.
Procedure: Laparoscopy — Veress needle was placed through the umbilicus and into the peritoneal cavity,After a pneumo-peritoneum has been achieved with a Veress needle, the primary trocar with sleeve (5mm in diameter) was placed at a similar angle in to the Veress needle

SUMMARY:
The hysteroscopy used was rigid continuous flow diagnostic hysteroscopy (Tuttligen, Karl Storz, Germany). It has a 30o panoramic optic which is 4mm in diameter and the diagnostic continuous flow outer sheath is 6.5 mm in diameter.

The patient was placed in lithotomy position with the buttocks projecting slightly beyond the table edge. A reflex camera (Olympus) with an objective that has a focal length varies from f70 to f140 together with (Karl Storz) special zoom length, adapter to Hopkins telescope and a suitable cableware used with computer flash unit. The hysteroscopic picture which appeared through the optic, transmitted on the monitor by the camera which is fitted on the eyepiece of the optic where the panoramic diagnostic hysteroscopy could be informed with better visualization and accuracy. The light generator which is a metal halide automatic light source with a 150 watt lamp (model G71A,Circon ACMI, Germany) was switched on and the high cable was attached to the hysteroscope. Dilatation of the cervix was avoided whenever possible to avoid leakage of the medium into the vagina. The hysteroscope was then introduced into the external os and advanced under vision along the axis of cervical canal.

Once the cavity was entered, an overview of the uterine cavity was performed. This was followed by systematic examination for fundus then tubal ostia on both sides then the uterine wall through slow rotatory movements of the telescope.

Diagnostic laparoscopy was done in the proliferative phase of the menstrual cycle .The patients were placed in the dorsal lithotomy position to allow vaginal access for uterine manipulation; the legs positioned so that the thighs are slightly flexed no more than 90o from the plane of the abdomen.

The patient was placed in the complete horizontal position, Veress needle was placed through the umbilicus and into the peritoneal cavity, the primary trocar with sleeve (5mm in diameter) was placed at a similar angle in to the Veress needle.

Secondary trocars were used, 2 secondary trocars were placed. The trocars were placed laterally, approximately 8 cm from the midline and 8 cm above the pubic symphysis to avoid the epigastric, vessels which are 5.5 cm from the midline at this level.

Then laparoscopic dye chromotubation was performed

DETAILED DESCRIPTION:
The hysteroscopy used was rigid continuous flow diagnostic hysteroscopy (Tuttligen, Karl Storz, Germany). It has a 30o panoramic optic which is 4mm in diameter and the diagnostic continuous flow outer sheath is 6.5 mm in diameter.

The patient was placed in lithotomy position with the buttocks projecting slightly beyond the table edge. The perineum and vagina were gently swabbed with povidone-iodine. The cervix was exposed was exposed with a posterior wall retractor and a tenaculum was applied to its anterior lip. The telescope was inserted into the sheath then flushed with distension media (saline) to expel any air. The technique used to provide uterine distension involved attaching plastic bags of saline to dual blood infusion tubing. Each bag was then wrapped in a pressure infusion cuff similar to that used to infuse blood under pressure with a pressure used 100mmHg. A reflex camera (Olympus) with an objective that has a focal length varies from f70 to f140 together with (Karl Storz) special zoom length, adapter to Hopkins telescope and a suitable cableware used with computer flash unit. The hysteroscopic picture which appeared through the optic, transmitted on the monitor by the camera which is fitted on the eyepiece of the optic where the panoramic diagnostic hysteroscopy could be informed with better visualization and accuracy. The light generator which is a metal halide automatic light source with a 150 watt lamp (model G71A,Circon ACMI, Germany) was switched on and the high cable was attached to the hysteroscope. Dilatation of the cervix was avoided whenever possible to avoid leakage of the medium into the vagina. The hysteroscope was then introduced into the external os and advanced under vision along the axis of cervical canal.

Once the cavity was entered, an overview of the uterine cavity was performed. This was followed by systematic examination for fundus then tubal ostia on both sides then the uterine wall through slow rotatory movements of the telescope.

Examination was considered normal if the endometrial cavity was easily distended by the medium with complete separation of its walls and vision of both tubal ostia.

Agglutination of the uterine walls or the presence of thick bands extending across the cavity or occlusion of ostial area or upper cavity indicated intrauterine adhesions (IUAs).

A longitudinal filling defect extending from the fundus downwards to a variable level indicated a uterine septum.

Any other pathological lesions such as polyps, submucous myomas were described according to their site, size and vascularity.

At the end of the procedure, the hysteroscope was slowly withdrawn through the cervical canal which was visualized to detect any lesion.

Diagnostic laparoscopy was done in the proliferative phase of the menstrual cycle .The patients were placed in the dorsal lithotomy position to allow vaginal access for uterine manipulation; the legs positioned so that the thighs are slightly flexed no more than 90o from the plane of the abdomen. The buttocks were slightly over the edge of the table but the sacrum was completely supported to the table, to avoid back strain. Once the primary trocar was placed, the patient was placed in no more than 25o Trendelenberg position to help keeping the bowel of the pelvis.

Clipping of the pubic hair was done, 3 - 4 cm above the symphysis pubis. Standard anti- septic preparation of the abdominal skin and the vagina were followed by placement of specially designed fenestrated laparoscopy drapes. Vaginal instruments were placed for uterine manipulation and then draped to keep the abdominal field separated from the lower vaginal field, followed by changing gloves, to avoid contamination of both the abdominal field and instruments placed into the abdominal cavity.

The patient was placed in the complete horizontal position, Veress needle was placed through the umbilicus and into the peritoneal cavity, avoiding both the retro peritoneal vessels and the intestinal tract. The abdominal wall was elevated by manually grasping the skin and the subcutaneous tissue to maximize the distance between the umbilicus and retroperitoneal vessels.

In persons of average weight, the lower anterior abdominal wall was grasped and elevated and the Veress needle was inserted toward the hollow of the sacrum at 45o angles. In patients who were obese, a more vertical approach, approximately 70-80o was required because of the increased thickness of the abdominal wall.

Correct placement of the Veress needle was confirmed by a number of methods, such as the hanging drop test, or injection and aspiration of fluid through the Veress needle. After a pneumo-peritoneum has been achieved with a Veress needle, the primary trocar with sleeve (5mm in diameter) was placed at a similar angle in to the Veress needle.

Secondary trocars were used, after identifying the epigastric vessels by transillumination and intraperitoneal observation, 2 secondary trocars were placed. The trocars were placed laterally, approximately 8 cm from the midline and 8 cm above the pubic symphysis to avoid the epigastric, vessels which are 5.5 cm from the midline at this level. Insertion of the trocar and removal of the sleeves were performed under direct laparoscopic visualization while observing for signs of hemorrhage. In case of bleeding, bipolar electro surgery was used to achieve hemostasis. Inspection of the whole peritoneal cavity, uterus, tubes ovaries, Douglas pouch, urinary bladder small and large intestine as well as the liver was done. Any abnormalities were noted and recorded.

Then laparoscopic dye chromotubation was performed to assess tubal patency bilaterally, by injecting methylene blue via the uterine catheter and observing spill through the fimbrial ends of the tubes. In case of negative spill, bluish discoloration and distention of the proximal parts of the tubes were noted.

At the end of the procedure, carbon dioxide inflation was stopped and the 2ry trocars were withdrawn under direct visualization, followed by deflation of the patient's peritoneal cavity and withdrawal of the 1ry trocars. Sutures were placed at the sites of 1ry and 2ry trocars to avoid incisional hernia.

ELIGIBILITY:
Inclusion Criteria:

1. Primary infertility defined as failure to conceive after one year of unprotected sexual intercourse
2. No detectable pelvic pathology based on history, physical examination and trans-vaginal ultrasound
3. Previous received treatment of six or more cycles in the form of ovulation stimulation
4. Normal HSG

Exclusion Criteria:

1. Couples with male factor infertility
2. Sexual problems
3. Contraindications to laparoscopy

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
tubal pathology | 6 months after hsterosalpingogram
  tubal patency tested through transcervical dye injection during laparoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No